CLINICAL TRIAL: NCT07162077
Title: The Effectiveness of Sodium Hypochlorite Application in Managing Opacities of Molar-incisor Hypomineralization on Incisors Using Resin Infiltration
Brief Title: Etch-bleach-seal Technique in Managing Opacities Related MIH Using Icon®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TishreenU- Pediatric Dentistry
Record Dates: First submitted 2025-08-26; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Molar Incisor Hypomineralisation
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: teeth will be randomized in two groups (test group and control group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium hypochlorite & ICON (Experimental): Resin infitration ( ICON (DMG, Hamburg, Germany)) and sodium hypochlorite 5.25%
  Interventions: Procedure: Sodium hypochlorite 5.25%
- ICON (Active Comparator): Resin infiltration ( ICON (DMG, Hamburg, Germany))
  Interventions: Procedure: ICON resin infiltration Material group in vivo

INTERVENTIONS:
Procedure: Sodium hypochlorite 5.25% — In the test group, the investigators will be applied sodium hypochlorite 5.25% by using cotton wad on the opacity before treatment, then after the first and second etching cycles (application of the Icon-Etch (ICON® -Etch; DMG, Hamburg, Germany) and Icon-dry (ICON® -Dry; DMG, Hamburg, Germany) according to the manufacturer's recommendations) as irrigation step and following the third -Etch etching cycle Icon-infiltrant (ICON® -Infiltrant; DMG, Hamburg, Germany) will be applied.
  Arms: Sodium hypochlorite & ICON
Procedure: ICON resin infiltration Material group in vivo — In control group, the investigators will be applied the same protocol of test group but without using sodium hypochlorite
  Arms: ICON

SUMMARY:
Objectives: to compare aesthetic effectiveness of resin infiltration with/without using sodium hypochlorite in managing opacities of MIH on incisors, and to compare parent's satisfaction with results of both application protocols.

Methods: Twenty-four teeth with yellow/ brown opacities of MIH, will be diagnosed according to EAPD diagnostic criteria, will be randomly allocated to test or control group. In the test group, the investigators will be applied sodium hypochlorite 5.25% by using cotton wad before treatment, then after the first and second etching cycles (application of the Icon-Etch (ICON® -Etch; DMG, Hamburg, Germany) and Icon-dry (ICON® -Dry; DMG, Hamburg, Germany) according to the manufacturer's recommendations) as irrigation step and following the third -Etch etching cycle Icon-infiltrant (ICON® -Infiltrant; DMG, Hamburg, Germany) will be applied . In control group, the investigators will be applied the same protocol of test group but without using sodium hypochlorite. The masking efficacy will be analyzed using the Lab System to calculate the color difference (ΔE) between the opacity and the adjacent enamel in Adobe Photoshop 2024. The infiltration proportion of opacity will be measured using Image J software and the infiltrated area will be expressed as a percentage. The satisfaction of the parents with the results of both application protocols will be compared using Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MIH-related opacities on the incisal and middle thirds of the buccal surface of their permanent incisors, ac- cording to EAPD diagnostic criteria of (MIH), only isolated lesions will be selected.

Exclusion Criteria:

* Teeth with resin composite restorations, previously treated by exter- nal bleaching, micro-abrasion or re-mineralization(fluoride varnish or calcium-based products such asCPP-ACP) will be excluded.
* Opacities present only on incisors without molar
* WSLs caused by orthodomtic treatment
* Teeth affected by dental fluorosis, Amelogenesis imperfecta and Tetracycline-pigmented teeth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Masking efficacy | The masking efficacy will be analyzed on day 1 and (7 - 10) days after day 1
  The masking efficacy will be analyzed using the Lab System to calculate the color difference (ΔE) between the opacity and the adjacent enamel in Adobe Photoshop 2024.

SECONDARY OUTCOMES:
The satisfaction of the parents | On day 1 and (7-10) days after
  Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- TishreenU, Latakia, Syria